CLINICAL TRIAL: NCT05033431
Title: An Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of a Single Dose of Brazikumab Administered by IV Infusion and SC Injection in Healthy Chinese and White Participants
Brief Title: Study to Evaluate the Pharmacokinetics (Movement of Drugs Within the Body), Safety and Tolerability of Brazikumab in Healthy Chinese and White Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D5271C00004
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants
Keywords: Inflammatory bowel disease; Brazikumab; Pharmacokinetics; Crohn's Disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 [Healthy Chinese Participants] (Experimental): Participants will receive a single intravenous (IV) infusion of brazikumab dose 1 on Day 1.
  Interventions: Drug: Brazikumab
- Group 2 [Healthy Chinese Participants] (Experimental): Participants will receive a single IV infusion of brazikumab dose 2 on Day 1.
  Interventions: Drug: Brazikumab
- Group 3 [Healthy Chinese Participants] (Experimental): Participants will receive a single subcutaneous (SC) injection of brazikumab dose 3 on Day 1.
  Interventions: Drug: Brazikumab
- Group 4 [Healthy Chinese Participants] (Experimental): Participants will receive a single SC injection of brazikumab dose 4 on Day 1.
  Interventions: Drug: Brazikumab
- Group 5 [healthy White participants] (Experimental): Participants will receive a single IV infusion of brazikumab dose 2 on Day 1.
  Interventions: Drug: Brazikumab
- Group 6 [healthy White participants] (Experimental): Participants will receive a single SC injection of brazikumab dose 4 on Day 1.
  Interventions: Drug: Brazikumab

INTERVENTIONS:
Drug: Brazikumab — Participants will receive IV or SC injection of brazikumab as per the group they are assigned.

SUMMARY:
This is a Phase I, single-centre, open-label, parallel-group, single dose study to evaluate the pharmacokinetics, safety and tolerability of Brazikumab in healthy male and female Chinese participants and healthy male and female White participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of giving signed and dated informed consent
* Healthy Chinese and White male and female participants aged 18 to 55 years (inclusive), at the time of signing the informed consent
* For White participants only:

  * Participant must be of European descent or White Latin American descent by participant report
* For Chinese participants only:

  * Participant was born in greater China, including Hong Kong, Macau, and Taiwan
  * Participant has 2 Chinese biological parents and 4 Chinese grandparents as confirmed by interview
  * Participant has not been living outside of greater China for more than 10 years at the time of the Screening period
* White male and female participants (Participant must be European descent or White Latin American descent)
* Participant who is overtly healthy as determined by medical evaluation
* Have a body mass index ≥ 18 kg/m^2 and ≤ 30 kg/m^2
* Female participants of childbearing potential must have a negative urine pregnancy test prior to administration of the investigational medicinal product (IMP) and must agree to use a highly effective method of birth control (confirmed by the Investigator) from enrolment throughout the study duration and for at least 18 weeks after last dose of the IMP
* Nonsterilised males who are sexually active with a female partner of childbearing potential should use protocol defined contraception method

Exclusion Criteria:

* History of any clinically significant disease or disorder in any body system
* Clinical signs and symptoms consistent with Coronavirus disease 2019 (COVID-19), eg, fever, dry cough, dyspnoea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to the Screening period or on admission
* History of alcohol or other substance abuse within the previous 5 years
* Known hypersensitivity to biologic therapy
* Taken any concomitant medications (including over-the-counter medications such as aspirin, acetaminophen, ibuprofen, herbal [including traditional Chinese medicinal products] or dietary supplements and cough syrup, as well as medicines requiring a prescription) within 14 days or 5 half-lives (whichever is longer), or St John's Wort within 30 days before the study drug administration
* Previously taken brazikumab or previously participated in an investigational study of brazikumab (previously known as AMG139 or MEDI2070)
* Participation in any other clinical investigation using an experimental drug within 30 days or 5 half-lives whichever is longer prior to dosing on Day 1
* For study participants for whom the COVID-19 vaccination is planned, vaccination (all doses) prior to first study drug dose may be advisable. If possible, the first dose of brazikumab should be given at least 30 days after the last dose of vaccine
* Blood or plasma donation within 60 or 30 days, prior to dosing on Day 1
* Any clinically significant abnormal findings in vital signs at the Screening period
* Abnormal electrocardiogram results thought to be clinically significant
* Abnormal and clinically significant results on physical examination, medical history, serum chemistry, haematology, or urinalysis
* Positive test results for anti-human immunodeficiency virus type 1 and type 2 antibodies, hepatitis B surface antigen and hepatitis B core antibody, anti-hepatitis C virus antibodies, human T-lymphotropic virus type 1 and human T-lymphotropic virus type 2 or tuberculosis at the Screening period
* Consumption of alcohol within 72 hours before administration of the study drug
* Positive test results for drug of abuse during the Screening period or on Day -1
* The participant has a condition or is in a situation which, in the Investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study
* Directly or indirectly involved in the conduct and administration of this study as an Investigator, Sub-investigator, study coordinator, or other study staff member; or employee of the Sponsor, or a first-degree family member, significant other, or relative residing with one of the above persons involved directly or indirectly in the study
* Female participant who is breastfeeding
* Evidence of a recent (within 6 months of Day 1) systemic fungal infection, requiring inpatient hospitalisation, and/or antifungal treatment
* Any infection requiring hospitalisation or treatment with IV anti-infectives (including anti-viral treatment) within 4 weeks prior to Screening
* Participant received a Bacille Calmette-Guérin vaccination within 12 months of Day 1 or any other live vaccine less than 4 weeks prior to Day 1 or is planning to receive any such vaccine over the course of the study
* Judgement by the Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements
* Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
* Participants who cannot communicate reliably with the Investigator

Detailed inclusion/exclusion criteria are in the study protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum (peak) drug concentration (Cmax) of brazikumab | Day 1 to Day 133
  Cmax of brazikumab in healthy Chinese and White participants will be evaluated.
Area under serum concentration-time curve from zero to infinity (AUCinf) of brazikumab | Day 1 to Day 133
  AUCinf of brazikumab in healthy Chinese and White participants will be evaluated.
Area under the serum concentration-time curve from zero to the last quantifiable concentration (AUClast) of brazikumab | Day 1 to Day 133
  AUClast of brazikumab in healthy Chinese and White participants will be evaluated.
Partial area under the serum concentration-time curve from time zero to 28 days postdose (AUC0-28d) of brazikumab | Day 1 to Day 133
  AUC0-28d of brazikumab in healthy Chinese and White participants will be evaluated.

SECONDARY OUTCOMES:
Number of participants with Adverse events (AEs) and Serious adverse events (SAEs) | From Screening period (Day -28 to Day -2) to Day 133 and Early termination visit
  Safety and tolerability of brazikumab in healthy Chinese and White participants will be evaluated.
Maximum observed serum (peak) drug concentration divided by the dose administered (Dose-normalised Cmax) of brazikumab | Day 1 to Day 133
  Dose-normalised Cmax of brazikumab in healthy Chinese and White participants will be evaluated.
Area under the plasma concentration-time curve from time zero to infinity divided by the dose administered (Dose-normalised AUCinf) of brazikumab | Day 1 to Day 133
  Dose-normalised AUCinf of brazikumab in healthy Chinese and White participants will be evaluated.
Area under the plasma concentration-time curve from time zero to the last quantifiable concentration divided by the dose administered (Dose-normalised AUClast) of brazikumab | Day 1 to Day 133
  Dose-normalised AUClast of brazikumab in healthy Chinese and White participants will be evaluated.
Partial area under the serum concentration-time curve from time zero to 28 days postdose divided by the dose administered (Dose-normalised AUC0-28d) of brazikumab | Day 1 to Day 133
  Dose-normalised AUC0-28d of brazikumab in healthy Chinese and White participants will be evaluated.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) of brazikumab | Day 1 to Day 133
  tmax of brazikumab in healthy Chinese and White participants will be evaluated.
Terminal elimination rate constant (λz) of brazikumab | Day 1 to Day 133
  λz of brazikumab in healthy Chinese and White participants will be evaluated.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) of brazikumab | Day 1 to Day 133
  t1/2λz of brazikumab in healthy Chinese and White participants will be evaluated.
Total body clearance of drug from serum after intravascular administration (CL) of brazikumab (IV only) | Day 1 to Day 133
  CL of brazikumab in healthy Chinese and White participants will be evaluated.
Volume of distribution following intravascular administration (based on terminal phase [Vz]) of brazikumab (IV only) | Day 1 to Day 133
  Vz of brazikumab in healthy Chinese and White participants will be evaluated.
Apparent total body clearance of drug from serum after extravascular administration CL/F of brazikumab (SC only) | Day 1 to Day 133
  CL/F of brazikumab in healthy Chinese and White participants will be evaluated.
Volume of distribution (apparent) following extravascular administration (based on terminal phase [Vz/F]) of brazikumab (SC only) | Day 1 to Day 133
  Vz/F of brazikumab in healthy Chinese and White participants will be evaluated.
Incidence of positive anti-drug antibodies to brazikumab in serum | Day 1 to Day 133
  Immunogenicity: incidence of brazikumab anti-drug antibodies in serum will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home